CLINICAL TRIAL: NCT01368939
Title: A Pilot, Single Centre, Prospective Clinical Study Investigation of the Acceptability of a Dedicated High Resolution Nuclear Breast Imaging Camera (MBI) in Breast Imaging of Patients Administered Tc-99m Sestamibi (ROSE)
Brief Title: Investigation of High Resolution Nuclear Breast Imaging Camera (MBI) in Patients Administered Tc-99m Sestamibi (ROSE)
Acronym: ROSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: HHSC-CPDC-001
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Breast Lesions
Keywords: breast imaging; MBI; dose reduction; Tc-99m; imaging; cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This research protocol is designed to evaluate a novel imaging camera, only one of three of it's kind in existence, in the diagnosis of breast cancer. The Molecular Breast Imaging Camera (MBI) is a gamma camera that images accumulation of 99mTc-Sestamibi, a radiopharmaceutical with high affinity for tissues of high cellularity and mitochondrial content; a common characteristic of breast cancers.

This camera represents a significant advancement over its predecessors as it has improved imaging geometry since it can be in direct contact with breast tissue and improved gamma photon detection capability through the use of cadmium zinc telluride (CZT) crystals (a semiconductor material) instead of NaI used in standard gamma cameras.

This project involves imaging patients with a baseline population risk of breast cancer, referred for myocardial perfusion imaging (MPI). This is possible because 99mTc-sestamibi is also used to image myocardial tissue. After the MPI study is performed to standard clinical specifications, the patient is simply imaged with the MBI.

The primary endpoint of this project is to assess acceptability of this imaging device by the patient through the use of a patient survey. Secondary endpoints are to correlate any findings on the MBI studies with standard breast imaging modalities including mammogram, ultrasound, and MRI. Image quality will be evaluated by the interpreting physicians. Also, in an effort to reduce radiation absorbed dose to the female breast, low injected dose images, obtained through post-processing by reframing acquired images, will be assessed for acceptable image quality and diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* females over 18 years of age
* completed a cardiac stress test using Tc-99m Sestamibi as the radiotracer prior to MBI imaging on the same day.
* signed consent form

Exclusion Criteria:

* pregnant or lactating
* history of invasive breast cancer or ductal carcinoma in situ
* prior bilateral mastectomy
* prior breast biopsy or surgery within 3 months
* any other conditions that based on the investigator's judgement, may impact the ability of the patient to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have completed a cardiac stress test with Tc-99m Sestamibi (same day) will be eligible for enrollment into the study. Females over the age of 18 and signed consent form. Subjects will be recruited from the cardiac care clinic on Site.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-09 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singnurkar, MD, FRCPC, Principal Investigator — HHSC, McMaster University, St. Joseph's Healthcare
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada